CLINICAL TRIAL: NCT00498797
Title: A Phase II, Double-blind, Placebo-controlled, Randomised Study to Assess the Efficacy and Safety of Docetaxel (Taxotere)/Prednisolone/ZD6474 vs Docetaxel/Prednisolone/Placebo in Patients With Hormone Refractory Prostrate Cancer (HRPC)
Brief Title: E3-Hormone Refractory Prostrate Cancer Taxotere Combination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D4200C00055; 2005-003593-16 (EudraCT Number)
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Results first posted 2011-05-24 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Prostate Cancer; Metastatic; Hormone Refractory
Keywords: prostate cancer; zactima; vandetanib; metastatic
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — vandetanib; Docetaxel; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Zactima (vandetanib)
Drug: Docetaxel
Drug: Prednisolone

SUMMARY:
The purpose of this study is to determine whether treatment with Zactima (vandetanib) in combination with Docetaxel and Prednisolone is more effective than the standard Docetaxel and Prednisolone alone for prostate cancer, in patients with Hormone refractory prostate cancer who have not previously received chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic hormone refractory prostate cancer defined as those patients with evidence of progression of disease in spite of castrate levels of testosterone indicated by rising levels of PSA
* No previous chemotherapy although those patients that have received estramustine can enter the study provided the estramustine was stopped 3 weeks before dosing of study drug
* screening PSA values >20ng/ml. this must be confirmed by two separate measurements at least 2 weeks apart

Exclusion Criteria:

* Treatment within 4 weeks before randomization and/or whilst on study, treatment with the following: 1)non-approved or experimental drug, 2)treatment with a drug with similar mechanism of action to ZD6474
* concurrent treatment with other anticancer agents, othr than docetaxel and prednisolone as defined in the protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2005-12; Primary Completion 2007-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (11):
- Brazil (2):
  - Research site, Rio de Janeiro
  - Research Site, São Paulo
- Germany (4):
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Kassel
  - Research Site, Tübingen
- Research Site, Budapest, Hungary
- South Africa (2):
  - Research Site, Bloemfontein
  - Research Site, Cape Town
- Sweden (2):
  - Research Site, Umeå
  - Research Site, Uppsala

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient randomised 24 January 2006, last patient randomised 24 Nov 2006, data cut off data 21 July 2007
Groups:
- Vandetanib: docetaxel/prednisolone/vandetanib
- Placebo: docetaxel/prednisolone/placebo
Period: Overall Study
Arm/Group | Vandetanib | Placebo
Started | 43 (randomised patients) | 43 (randomised patients)
Completed | 5 (ongoing study treatment at data cut-off) | 14 (ongoing study treatment at data cut-off)
Not Completed | 38 | 29
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Adverse Event | 12 | 5
Not completed — Condition under investigation worsened | 19 | 21
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vandetanib | Placebo | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Continuous [Mean (Full Range); unit: years] | 67 [47 to 81] | 67 [43 to 79] | 67 [43 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 43 | 43 | 86

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen (PSA) Response
Description: Prostate Specific Antigen (PSA) response was defined as a reduction of at least 50% from baseline at any assessment, confirmed by a second assessment 2-4 weeks after the initial response
Time Frame: PSA measurements were to be performed at screening, at baseline (>2 weeks after screening) and every 3 weeks during the study. Any response was to be confirmed 2-4 weeks after the initial assessment of a 50% fall in PSA from baseline
Measure: Number; unit: Participants
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 43 | 43
Participants | 17 | 29

2. Secondary Outcome: Number of Patients With an Objective Disease Progression Event
Description: Number of patients with objective disease progression or death (by any cause in the absence of objective progression)
Time Frame: RECIST tumour assessments carried out at screening and then as per site clinical practice until objective progression. The only additional mandatory tumour assessment visit is at the point of data cut-off (21 July 2007 or up to 7 days in advance of DCO)
Measure: Number; unit: Participants
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 43 | 43
Participants | 28 | 26

ADVERSE EVENTS:
Arm/Group | Vandetanib | Placebo
Serious Adverse Events (participants affected / at risk) | 23/43 | 15/43
Other Adverse Events (participants affected / at risk) | 38/43 | 39/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib (N=43) | Placebo (N=43)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 1
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 1
BLINDNESS (Eye disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 1
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 1
FATIGUE (General disorders) | 0 | 1
PYREXIA (General disorders) | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 3 | 1
DIVERTICULITIS (Infections and infestations) | 1 | 0
LOBAR PNEUMONIA (Infections and infestations) | 1 | 0
PERIRECTAL ABSCESS (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
EPILEPSY (Nervous system disorders) | 1 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 1 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 | 1
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 1 | 0
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 | 0
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
THROMBOPHLEBITIS (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib (N=43) | Placebo (N=43)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 5
NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 4
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 3
PALPITATIONS (Cardiac disorders) | 3 | 0
VERTIGO (Ear and labyrinth disorders) | 3 | 1
LACRIMATION INCREASED (Eye disorders) | 4 | 7
CONJUNCTIVITIS (Eye disorders) | 1 | 3
NAUSEA (Gastrointestinal disorders) | 7 | 16
DIARRHOEA (Gastrointestinal disorders) | 10 | 13
CONSTIPATION (Gastrointestinal disorders) | 4 | 10
VOMITING (Gastrointestinal disorders) | 1 | 7
STOMATITIS (Gastrointestinal disorders) | 4 | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 3
DYSPEPSIA (Gastrointestinal disorders) | 3 | 3
FATIGUE (General disorders) | 16 | 14
ASTHENIA (General disorders) | 5 | 7
OEDEMA PERIPHERAL (General disorders) | 4 | 7
PYREXIA (General disorders) | 1 | 4
CHILLS (General disorders) | 3 | 1
NASOPHARYNGITIS (Infections and infestations) | 4 | 6
URINARY TRACT INFECTION (Infections and infestations) | 5 | 3
BRONCHITIS (Infections and infestations) | 0 | 3
ANOREXIA (Metabolism and nutrition disorders) | 4 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 6
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 5
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3 | 4
DYSGEUSIA (Nervous system disorders) | 8 | 5
HEADACHE (Nervous system disorders) | 1 | 5
DIZZINESS (Nervous system disorders) | 3 | 3
HYPOAESTHESIA (Nervous system disorders) | 0 | 3
PARAESTHESIA (Nervous system disorders) | 1 | 3
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 3 | 2
INSOMNIA (Psychiatric disorders) | 8 | 7
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 4
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 | 1
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 3 | 1
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 3
ALOPECIA (Skin and subcutaneous tissue disorders) | 16 | 19
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 5 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 4 | 1
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 4 | 1
ONYCHOMADESIS (Skin and subcutaneous tissue disorders) | 3 | 1
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 3 | 2
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 3 | 0
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 3 | 1
HYPERTENSION (Vascular disorders) | 6 | 1
FLUSHING (Vascular disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.